CLINICAL TRIAL: NCT07117773
Title: Changes in Hydration Status of PepsiCo Frontline Workers in a Manufacturing Facility Over the Course of Multiple Shifts
Status: Completed | Type: Observational
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Other Study IDs: PEP-2509
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Hydration Status
Keywords: hydration; ergonomics; industrial worker; observational

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: PepsiCo Frontline Workers

SUMMARY:
Physically demanding occupations (PDO) require high levels of energy expenditure, mental acuity, and technical skills. Sometimes this work is performed in extreme environments during hot/humid summer months. Previous research shows that dehydration and heat stress can increase risk of heat-related illness, reduced cognitive function, and work capacity. While this impact of physically demanding work in extreme environmental conditions is often studied in firefighters, military personnel, and athletes, and even agricultural workers, manufacturing and warehouse workers ("the industrial athlete") are underrepresented in the literature.

The purpose of the study is to examine the impact hydration status of the industrial athlete (i.e., frontline manufacturing and warehouse workers at PepsiCo facilities) prior to, during, and after their shift over a typical work week has on work performance.

Note: Recruitment is limited to PepsiCo Frontline Employees Only. Do not contact study official for enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as a healthy male or female
* Subject is 18-65 years of age
* The subject is currently employed by PepsiCo at a bottling facility
* Subject can read and comprehend English
* Subject has worked for PepsiCo for 2 months or longer
* Willing to agree with what is outlined in the informed consent form.

Exclusion Criteria:

* Subject has an allergy to adhesives
* Female subject is pregnant or nursing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Frontline manufacturing and warehouse workers at Orlando PBNA Bottling Facility
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2025-08-08 (Actual); Primary Completion 2025-08-22 (Actual); Study Completion 2025-08-24 (Actual)

PRIMARY OUTCOMES:
Acute Urine Specific Gravity | Post-shift USG compared to pre-shift USG (8-12 hours from baseline) on consecutive test day 1-4 over calendar week.
  USG digital pen refractometer (au)
Chronic Urine Specific Gravity | pre- and post- 8-12 hour shift USG on the last test day compared to pre- and post-8-12 hour shift USGs at baseline. Over 4 consecutive test days during a calendar week.
  Digital pen refractometer (au)

SECONDARY OUTCOMES:
Urine Color | 15 minutes pre- 9-12 hour shift and 15 minutes post- 8-12 hour shift, consecutive test day 1-4 over a calendar week.
  1=most dilute to 7= least dilute
Body Weight | 15 minute pre- 8-12 hour shift on the first test day
  (kg)
Sweat Loss | over the course of an 8-12 hour shift, consecutive test day 2-4 over a calendar week.
  (mL) monitored using the Epicore Connected Hydration device
Sweat Rate | over the course of an 8-12 hour shift, consecutive test day 2-4 over a calendar week.
  (mL/hr) monitored using the Epicore Connected Hydration device
Sodium Concentrations | over the course of an 8-12 hour shift, consecutive test day 2-4 over a calendar week.
  (g/L) monitored using the Epicore Connected Hydration device
Sodium Loss | over the course of an 8-12 hour shift, consecutive test day 2-4 over a calendar week.
  (g) monitored using the Epicore Connected Hydration device
Fluid Intake | Each time water bottle is refilled over 8-12 hour shift, consecutive test day 1-4 over a calendar week.
  (g) pre-shift bottle weight before and after filled with water compared to pre- and post-refill bottle weight.
Measurment of physical activity and movement (Accelerometry) | over the course of an 8-12 hour shift, consecutive test day 2-4 over a calendar week.
  Assessed using the LifeBooster Senz devices. Device measures frequency and severity of movements and posture.
work-to-rest ratio | over the course of an 8-12 hour shift, consecutive test day 2-4 over a calendar week.
  Assessed using the LifeBooster Senz devices. Device measures frequency and severity of movements and posture.
Mental and Physical Energy and Fatigue | 30 minutes pre- and 30 minutes post- 8-12 hour shift on consecutive test day 1-4, over a calendar week
  Visual Analog Scale (VAS): 6 questions to describe capacity for physical activity anchored from No to Strongest Feelings and 6 questions describe capacity for mental activity anchored from No to Strongest Feelings.
Thirst | 30 minutes pre- and 30 minutes post- 8-12 hour shift on consecutive test day 1-4, over a calendar week
  Visual Analog Scale- 6 questions: 4 questions are anchored from not at all or none to very, and 2 questions are anchored from pleasant to unpleasant.
Prior Night Sleep Quality | 30 minutes pre- 8-12 hour shift on consecutive test day 1-4, over a calendar week
  Pittsburgh Sleep Quality Index (PSQI). Measures sleep quality through seven areas: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction over the last month. Score of the PSQI ranges from 0 to 3, with 3 indicating the greatest dysfunction or disturbance. The seven component scores are then summed to obtain a global PSQI score, which ranges from 0 to 21. Higher scores indicate poorer sleep quality, with a score greater than 5 suggesting significant sleep difficulties

CONTACTS AND LOCATIONS:
Overall Officials: Philip Agostinelli, PhD, Principal Investigator — PepsiCo R&D/Gatorade and Sports Science Institute
Locations (1):
- Gatorade Sports Science Institute, Bradenton, Florida, United States

IPD SHARING:
Plan to Share IPD: No